CLINICAL TRIAL: NCT02346877
Title: A Multicenter, Historical Control Study to Evaluate the Effects of Personalized Patient Counselling on Persistence to Enbrel® Therapy in Subjects With Rheumatoid Arthritis (PerSuit)
Brief Title: Evaluate Effects of Personalized Patient Counselling for Enbrel® Therapy in Adults With Rheumatoid Arthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20130340
Record Dates: First submitted 2015-01-07; First posted 2015-01-27 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Persistence to Enbrel
Keywords: Enbrel; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care Cohort (No Intervention): The first 100 participants will be enrolled in the standard of care (control) cohort. These participants will receive treatment with Enbrel® (etanercept) in routine clinical practice and will complete a 52 week study period as per the investigator's standard of care.
- Personalized Patient Counselling Cohort (Other): Initiation of the personalized patient counselling cohort will begin after 75% of participants in the control cohort have been analyzed and shown not to have high persistence. Participants will receive Enbrel® (etanercept) therapy in routine clinical practice and personalized patient counselling based on the Information-Motivation-Strategy (IMS) model based on Beliefs about Medicines Questionnaire (BMQ) baseline results through a patient assistance program for patients on Enbrel (etanercept) therapy.
  Interventions: Behavioral: Personalized Patient Counselling

INTERVENTIONS:
Behavioral: Personalized Patient Counselling — In the interventional cohort participants enrolled on the study will receive personalized patient counselling using the IMS-model based on the baseline BMQ results through a patient assistance program for patients on Enbrel (Etanercept) therapy.
  Arms: Personalized Patient Counselling Cohort

SUMMARY:
This study will evaluate whether the effect of personalized patient counselling tool, Information-Motivation-Strategy (IMS) based on the results of the Beliefs about Medicines Questionnaire (BMQ) will improve persistence of Enbrel (etanercept) therapy at week 52 in subjects with rheumatoid arthritis over the historical control as estimated by the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent prior to any study specific procedures
* diagnosed with rheumatoid arthritis and eligible for treatment with Enbrel® (etanercept)
* Subject has been prescribed and has access to commercial Enbrel® (etanercept) (50mg once weekly) according to the subject's health insurance
* Completion of all required safety assessments before starting treatment with Enbrel® (etanercept)

Other Inclusion Criteria May apply.

Exclusion Criteria:

* previously received treatment with a biologic disease modifying antirheumatic drug (DMARD) and/or Tofacitinib.
* Malignancy (except nonmelanoma skin cancers, cervical or breast ductal carcinoma in situ) within the last 5 years
* refusal to consent to enroll in the Enliven program
* Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s)

Other Exclusion Criteria May Apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (14):
- Canada (14):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Fredericton, New Brunswick
  - Research Site, Quispamsis, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Trois-Rivières, Quebec

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated at 15 centers in Canada, of which 8 centers enrolled participants. The first participant was enrolled on 14 April 2015 and the last participant enrolled on 13 October 2015.
Pre-assignment Details: Eligible participants were to be enrolled in the standard of care (control) cohort and complete the 52-week study period. Data from 75% of the group were to be analyzed before enrolling participants in the interventional cohort. As the study was prematurely closed due to slow enrollment, the interventional cohort was not enrolled.
Groups:
- Standard of Care (Control) Cohort: The first 100 participants were to be enrolled in the standard of care cohort. These participants received treatment with Enbrel® (etanercept) in routine clinical practice and were to complete a 52 week study period as per the investigator's standard of care.
- Personalized Patient Counselling (Interventional) Cohort: Participants enrolled in the interventional cohort were to receive Enbrel® (etanercept) therapy and personalized patient counselling using the Information-Motivation-Strategy (IMS) model based on Beliefs about Medicines Questionnaire (BMQ) results through a patient assistance program for patients on Enbrel (etanercept) therapy.
Period: Overall Study
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort
Started | 19 | 0
Completed | 0 | 0
Not Completed | 19 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Administrative Decision | 1 | 0
Not completed — Sponsor Decision | 12 | 0
Not completed — Missing | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort | Total
Number analyzed (Participants) | 19 | 0 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (10.1) |  | 57.1 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 |  | 14
  Male | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Persistence of Study Drug Measured at 52 Weeks
Description: A participant is persistent if the date of the last prescription filled plus the number of weeks supply of the prescription is greater than or equal to 52 weeks from enrolment and the eDiary confirms Enbrel® from the prescription was injected. A participant is not persistent if the last prescription filled plus the number of weeks supply of the prescription is less than 52 weeks from enrolment and the eDiary confirms there was no injection of Enbrel®, or, a participant is not persistent if the participant has a gap in treatment of more than 4 consecutive weeks for no medical reason at any time in the 52 week study period.
Time Frame: 52 weeks
Population: Efficacy endpoints were not evaluated because the study was prematurely closed and no participants completed the study.
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Adherence to Study Drug up to 52 Weeks
Description: A participant's adherence is determined as a medication possession ratio (MPR) of at least 80%. The MPR is the ratio of the total number of weeks' supply, based on pharmacy data, of Enbrel® divided by either 52 weeks or duration on study if a physician stops prescribing Enbrel® due to an adverse drug reaction or lack of efficacy.
Time Frame: 52 weeks
Population: Efficacy endpoints were not evaluated because the study was prematurely closed and no participants completed the study.
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Beliefs About Medicines Questionnaire (BMQ)
Description: BMQ consists of two five-item scales assessing patients' beliefs about the necessity of Enbrel® for controlling their rheumatoid arthritis and their concerns about potential adverse consequences of taking Enbrel®. Using a five-point Likert scale, on each of necessity and concerns, the individual items within both scales are summed. The total scores for the Necessity and Concerns Scales range from 5 to 25. Higher scores indicate stronger beliefs.
Time Frame: 52 weeks
Population: Efficacy endpoints were not evaluated because the study was prematurely closed and no participants completed the study.
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Only adverse drug reactions and serious adverse drug reactions were collected in this study.
Arm/Group | Standard of Care (Control) Cohort | Personalized Patient Counselling (Interventional) Cohort
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/0
Other Adverse Events (participants affected / at risk) | 1/19 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care (Control) Cohort (N=19) | Personalized Patient Counselling (Interventional) Cohort (N=0)
Injection site reaction (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.